CLINICAL TRIAL: NCT02389634
Title: Identification of Novel Molecular Markers for Vasospasm From the Cerebrospinal Fluid (CSF) of Patients With Aneurysmal Subarachnoid Hemorrhage
Brief Title: Identification of Novel Molecular Markers for Vasospasm
Status: Completed | Type: Observational
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Translational Genomics Research Institute (Other)
Responsible Party: Principal Investigator, Lori Wood, Research Operations Manager, St. Joseph's Hospital and Medical Center, Phoenix
Other Study IDs: 10BN048
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Vasospasm; Subarachnoid Hemorrhage
MeSH Terms: conditions — Vasospasm, Intracranial; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and cerebrospinal fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to identify novel genetic and protein markers for the process of cerebral vasospasm following aneurysmal subarachnoid hemorrhage.

DETAILED DESCRIPTION:
Cerebral vasospasm is a recognized and poorly understood complication for many patients who have aneurysmal subarachnoid hemorrhage. Constriction of the cerebral arterial vasculature occurs as free subarachnoid blood under high pressure comes into contact with the surfaces of vessels, particularly in the basal cisterns. However, the exact pathophysiology of vasospasm is unknown. Morbidity and mortality rates for vasospasm are high despite improvements in management. Excluding the initial hemorrhage, cerebral vasospasm is recognized as the main cause of substantial disability and death. Cerebral vasospasm kills 7% of patients, and causes severe deficit in another 7%. Cerebral vasospasm almost never occurs before day 3, has maximal incidence at days 6-8, and rarely occurs after day 17. The disorder is clinically characterized by confusion or decreased consciousness with focal neurological deficit.

Experimental evidence suggests that red blood cell hemolysis and subsequent release of oxygen, hemoglobin, reactive oxygen species, and other as yet undescribed mediators are necessary for the development of vasospasm. The goal of this study is to use modern tools of genomics to identify novel molecular markers for the process of vasospasm by studying the release of micro ribonucleic acids (RNA) that are secreted into the cerebrospinal fluid following the initiation of vasospastic cascades. Micro RNA's have recently been identified as important regulators of many cellular processes including cell cycle progression, proliferation, tumor suppressors, oncogenes, and regulators of metabolic pathways. The researchers propose to study the levels of annotated micro RNA's in the cerebrospinal fluid (CSF) of patients who present with subarachnoid hemorrhage from presentation through the hospital stay. The researchers will correlate the level of these micro RNA's with patient clinical presentation, including transcranial Doppler measurements, Glasgow Coma Scale score, vital signs, and angiographic studies. It is well established that the process of vasospasm occurs over the course of many days. Long before vasospasm becomes clinically evident, cellular processes causing spasm are in action and the researchers hope to identify micro RNA mediators of these processes using high throughput screening methods.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with aneurysmal subarachnoid hemorrhage within 24-hours of bleed.
* Receive either open vascular clipping or endovascular coiling.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients arriving at the hospital >24-hours post-hemorrhage.
* Patients who are not candidates for further care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with aneurysmal subarachnoid hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Identification of vasospasm via microRNA mediators prior to clinically evident signs and symptoms | 30 days
  Identification of vasospasm via microRNA mediators prior to clinically evident signs and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Spetzler, MD, Principal Investigator — Saint Joseph's Hospital and Medical Center/Barrow Neurological Institute
Locations (1):
- Barrow Neurological Institute at St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided